CLINICAL TRIAL: NCT05434520
Title: Relieving the Bile Ducts Prior to Pancreatoduodenectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Waqas Farooqui, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: PDPTC1
Record Dates: First submitted 2022-05-28; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pancreas Cancer; Surgery-Complications; Biliary Fistula
Keywords: pancreatoduodenectomy; complications; percutaneous transhepatic biliary drainage
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative biliary drainage: Patients who had undergone preoperative biliary drainage (ERC og PTC) prior to pancreatoduodenectomy
  Interventions: Procedure: Preoperative biliary drainage (ERC og PTC-aided)
- No preoperative biliary drainage: Patients who had not undergone preoperative biliary drainage (ERC og PTC) prior to pancreatoduodenectomy

INTERVENTIONS:
Procedure: Preoperative biliary drainage (ERC og PTC-aided) — Placement of biliary stent (plastic, covered SEMS, uncovered SEMS) endoscopic by ERC or placement of plastic catheter by PTC
  Groups: Preoperative biliary drainage

SUMMARY:
The aim of this study was to assess the risk and complications after preoperative drainage of biliary obstruction in patients who underwent pancreatoduodenectomy.

A retrospective cohort study of all patients who underwent pancreatoduodenectomy from January 1st, 2015 to September 30th, 2021. Patients who had preoperative bile duct drainage were compared to patients without intervention. Type of interventions, complications and outcome after surgery were compared using univariate and multivariate analysis.

DETAILED DESCRIPTION:
Obstructive jaundice is a common problem in pancreatic and periampullary tumors, but preoperative biliary drainage in patients with hyperbilirubinemia is still controversial. The aim of this retrospective cohort study was to assess the risk and complications after preoperative drainage of biliary obstruction in patients who underwent pancreatoduodenectomy.

A retrospective cohort study of all patients who underwent pancreatoduodenectomy from January 1st, 2015 to September 30th, 2021.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had undergone pancreatoduodenectomy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who had undergone pancreatoduodenectomy from January 1st, 2015 to September 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Post-operative complication score (Clavien-Dindo) | During hospital admission, median time 13 days, up to 390 days.
  The prevalence of complications graded according to Clavien-Dindo score after pancreatoduodenectomy. Clavien-Dindo 0 is no complications, Clavien-Dindo 5 means complications resulting in mortality.
30-day Mortality | up to 30 days
  30-day mortality rate post-pancreatoduodenectomy
90-day Mortality | up to 90 days
  90-day mortality rate post-pancreatoduodenectomy
Length of Hospital Stay | Days from admission until discharge, up to 390 days, median time 13 days
  Accumulated length of hospital stay from the admission day prior to pancreatoduodenectomy, till the day of discharge.
30-day Readmission | up to 30-days from hospital discharge
  Prevalence of readmission within 30-days after discharge following pancreatoduodenectomy.

SECONDARY OUTCOMES:
Complications following preoperative bile duct drainage | up to 7 days after bile duct drainage
  Prevalence of cholangitis, pancreatitis, iatrogenic perforation, post-procedural bleeding and post-procedural thrombosis
Time from Bile Duct Drainage to Pancreatoduodenectomy | Days from bile duct decompression to pancreatoduodenectomy, median time 32 days, up to 534 days
  Time from Bile Duct Decompression to pancreatoduodenectomy.
Histological Specimen | Obtained within 21 days after resection
  Histological diagnosis of the resection specimens divided in malignant (ductal adenocarcinoma, cholangiocarcinoma, papillary carcinoma, duodenal adenocarcinoma, neuroendocrine tumor, other pancreatic carcinoma, other malignancy in the pancreas) and benign (IPMN, other benign diseases).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capitol, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and/or analyzed during the current study are not publicly available due to a restriction agreement with the Danish Data Protection Agency but are available from the corresponding author on reasonable request.